CLINICAL TRIAL: NCT07098715
Title: Closure Of Cryptoglandular Fistula-in-ano And Associated Non-healing Draining Wounds With Kerecis SurgiClose
Brief Title: A Study Of Cryptoglandular Fistula-in-ano And Associated Non-healing Draining Wounds With Kerecis SurgiClose
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicholas P. McKenna, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-007753
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fistula-in-ano; Draining Wound
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intact Kerecis Fish Skin (Experimental): To assess shot-term outcomes (rates of healing) using Kerecis intact fish skin to heal cryptoglandular fistula-in-ano and associated chronic non-healing draining wounds.
  Interventions: Device: Kerecis fish skin

INTERVENTIONS:
Device: Kerecis fish skin — To assess shot-term outcomes (rates of healing) using Kerecis intact fish skin to heal cryptoglandular fistula-in-ano and associated chronic non-healing draining wounds.

SUMMARY:
The purpose of this study is to determine feasibility of Kerecis intact fish skin for healing of fistula-in-ano and associated non-healing draining wounds.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ≥18 years old
* Cryptoglandular fistula-in-ano (primary or recurrent)
* The ability to give appropriate consent

Exclusion Criteria:

* Age <18 years old
* Pregnant (as determined by urine test)
* Any known allergies or sensitivities to fish material
* Prisoners
* Inflammatory bowel disease
* Fistula-in-ano associated with:

  * Anal cancer
  * Rectal cancer
  * Extramammary Paget's disease
  * Hidradenitis suppurativa
  * Anal condyloma
  * Active infection / abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Fistula healing | From device implant until 6 months after
  Assess healing of the fistula. This will be determined based on physical examination. A healed fistula will be a patient who 6 months after surgery no longer has drainage or evidence of infection. The internal opening should be closed on physical exam. The internal opening should feel closed on digital rectal exam. This will be assessed in each patient to determine the overall rate of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas P. McKenna, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials